CLINICAL TRIAL: NCT06829602
Title: PREnatal Syphilis Point-of-care ScreenING in an Urban Low-barrier Clinic: A Prospective Single Arm Feasibility Trial
Brief Title: The Feasibility of Implementing Syphilis Point-of-care Testing Into a Prenatal Clinic for People Facing Barriers to Care
Acronym: PRESSING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AS1-192615
Record Dates: First submitted 2025-01-05; First posted 2025-02-17 (Actual); Last update posted 2025-07-06 (Actual); Status verified 2025-06

CONDITIONS: Syphilis
Keywords: syphilis; pregnancy; access to care; acceptability; point-of-care test
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation of syphilis/HIV point-of-care testing (Experimental): The syphilis/HIV point-of-care test will be offered to all prenatal clients with at least 1 risk factor for syphilis, and to the sexual partners of syphilis-positive participants
  Interventions: Diagnostic Test: Rapid Syphilis/HIV point-of-care test

INTERVENTIONS:
Diagnostic Test: Rapid Syphilis/HIV point-of-care test — The INSTI Multiplex HIV/Syphilis Duo Antibody Test is a rapid immunoassay that can detect HIV and syphilis antibodies in the blood using finger-prick blood samples. The test is Health Canada-approved.

SUMMARY:
The goal of this clinical trial is to learn if a finger-prick blood test for rapid diagnosis of syphilis infection can be implemented in a low-barrier prenatal clinic for people at risk of syphilis in pregnancy. The test gives results in 5 minutes and also tests for HIV.

The main questions the study aims to answer are:

* How often do pregnant people at risk of syphilis agree to the rapid test?
* How well do healthcare providers perform the rapid test?
* Does the rapid test speed up diagnosis and treatment of syphilis in pregnant people and their sexual partners?

Participants will:

* Give feedback about why they did or did not want to take the rapid test, and what their experience was taking the test; and
* Share information about their health, pregnancy, and syphilis treatment (if applicable).

DETAILED DESCRIPTION:
Early testing and treatment for syphilis during pregnancy, along with treating sexual partners, can prevent infection of the baby (known as congenital syphilis). However, many pregnant people at risk of syphilis also face barriers to prenatal care due to social determinants of health such as substance use and unstable housing. These barriers may lead to delays in management of syphilis in pregnancy, which may result in poor maternal and infant health outcomes.

A major issue is the standard syphilis blood test. This test takes about a week to return results. This delay makes it difficult to communicate positive results to people with limited phone or internet access, and it can be hard for people to return for treatment. Additionally, it may be challenging to take blood for the syphilis test from people whose veins are damaged from intravenous drug use. As a result, syphilis diagnosis and/or treatment in pregnancy may be delayed or missed altogether.

Health Canada has approved a point-of-care test for syphilis and HIV that uses a finger-prick blood sample and gives results in 5 minutes. This rapid test enables same-day syphilis treatment initiation with intramuscular penicillin antibiotic, and could overcome some of the barriers described above. However, point-of-care syphilis testing has not been studied in pregnant people facing barriers to prenatal care.

An urban low-barrier prenatal clinic (Maternity Centre of Hamilton) will implement the point-of-care syphilis/HIV test as part of regular care. The test will be offered to pregnant clients at risk of syphilis, and to the sexual partners of syphilis-positive pregnant clients, given the critical importance of treating partners to prevent re-infection during pregnancy. Over 1 year, the study will evaluate the feasibility of test implementation, in terms of acceptability by clients and test performance by clinicians. The study will also preliminarily assess whether the point-of-care test improves timeliness and adequacy of treatment of syphilis-positive pregnant clients and their sexual partners. The investigators did not feel it was ethical to have a control group with delayed access to point-of-care testing given the potential harms of delayed diagnosis of syphilis in pregnancy; rather, baseline data regarding management of syphilis in pregnancy at the clinic will be established using retrospective chart review, and compared to syphilis management over the study period.

Importantly, if pregnant clients or sexual partners decline study participation, they are still eligible for point-of-care testing to learn their syphilis and HIV status.

ELIGIBILITY:
1. Pregnant people

   Inclusion Criteria:
   * Pregnant clients with at least one risk factor for syphilis infection:

     1. Substance use or accessed addiction services in the past 1 year
     2. Unstable housing in the past 1 year
     3. Multiple sexual partners in the past 1 year
     4. History of a sexually transmitted or blood-borne infection (STBBI)
     5. Late to prenatal care (initial prenatal visit >20 weeks)
   * Eligible for syphilis screening at that clinic visit, as per Public Health guidelines

   Exclusion Criteria:
   * Previous syphilis diagnosis
   * Not competent to consent to study participation
2. Sexual partners

Inclusion Criteria:

* Sexual partners of pregnant clients who are newly diagnosed with syphilis
* Physically present in the clinic

Exclusion Criteria:

* Previous syphilis diagnosis
* Not competent to consent to study participation

Ages: 13 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 77 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of pregnant clients with syphilis risk factors who undergo syphilis/HIV point-of-care testing the first time it is offered | Single time-point - At time of first offer of point-of-care test - approximately 5 minutes

SECONDARY OUTCOMES:
Proportion of pregnant participants with syphilis risk factors who undergo syphilis/HIV point-of-care testing at least once during pregnancy | From the first prenatal clinic visit until the end of pregnancy - up to 8 months
Proportion of pregnant participants who undergo syphilis/HIV point-of-care testing, and are willing to undergo the test in future based on post-test survey | Single time-point - at time of post-test survey - approximately 5 minutes
Proportion of partner participants who undergo syphilis/HIV point-of-care testing, and are willing to undergo the test in future based on post-test survey | Single time-point - at time of post-test survey - approximately 5 minutes
Proportion of syphilis/HIV point-of-care tests with valid results on clinician's first attempt, as defined by the manufacturer's instructions | From initiation to completion of point-of-care test - approximately 5 minutes
Proportion of syphilis/HIV point-of-care tests that are correctly interpreted by the clinician, as per consensus of 2 blinded independent study staff reviewing digital photographs of the results | From initiation to completion of point-of-care test - approximately 5 minutes
Proportion of pregnant participants with a positive syphilis point-of-care test, who receive same-day treatment initiation with penicillin | From positive syphilis point-of-care test result until end of clinic visit - up to 3 hours
Time to communicate test results to syphilis serology-positive pregnant participants, from date of first positive syphilis test (days) | From the day of syphilis testing to notification of client - range 5 minutes to 8 months
Time to first penicillin treatment for syphilis serology-positive pregnant participants, from date of first positive syphilis test (days) | From the day of syphilis testing to treatment of client - range 5 minutes to 8 months
Proportion of syphilis serology-positive pregnant participants who receive any syphilis treatment in pregnancy | From the day of syphilis testing to end of pregnancy - up to 8 months
Proportion of syphilis serology-positive pregnant participants who receive the recommended treatment in pregnancy, based on syphilis staging | From the day of syphilis testing to treatment of client - up to 8 months
Time to first penicillin treatment of partner participants, from date of pregnant person's date of first positive syphilis test (days) | From the day of pregnant person's syphilis testing to treatment of partner - range 1 hour to 8 months
Proportion of partner participants who receive any syphilis treatment during pregnancy | From the day of pregnant person's syphilis testing to treatment of partner - up to 8 months
Proportion of partner participants who receive the recommended syphilis treatment during pregnancy, based on their syphilis staging | From the day of pregnant person's syphilis testing to treatment of partner - up to 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura K Erdman, MD PhD FRCPC, Principal Investigator — McMaster University
Locations (1):
- Maternity Centre of Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No